CLINICAL TRIAL: NCT04266912
Title: DNA Damage Repair (DDR) Inhibitor-Based Basket of Baskets Phase I/II Trial in Patients With Advanced Solid Tumors Harboring Aberrations in DDR Genes (D-BoB)
Brief Title: Avelumab and M6620 for the Treatment of DDR Deficient Metastatic or Unresectable Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-1059; NCI-2019-07598 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-1059 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-11-26; First posted 2020-02-12 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Malignant Solid Neoplasm; Refractory Malignant Solid Neoplasm; Unresectable Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — avelumab; berzosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Escalation Dose Level 1 (Experimental): Berzosertib 240 mg/m2 once weekly + Avelumab 800 mg IV on days 1 and 15 of each 28-day cycle
  Interventions: Drug: Avelumab; Drug: Berzosertib
- Escalation Dose Level 2 (Experimental): Berzosertib 480 mg/m2 once weekly + Avelumab 800 mg IV on days 1 and 15 of each 28-day cycle
  Interventions: Drug: Avelumab; Drug: Berzosertib
- Expansion Dose Level 1 (Experimental): Berzosertib 240 mg/m2 once weekly + Avelumab 800 mg IV on days 1 and 15 of each 28-day cycle
  Interventions: Drug: Avelumab; Drug: Berzosertib
- Expansion Dose Level 2 (Experimental): Berzosertib 480 mg/m2 once weekly + Avelumab 800 mg IV on days 1 and 15 of each 28-day cycle
  Interventions: Drug: Avelumab; Drug: Berzosertib

INTERVENTIONS:
Drug: Avelumab — Given IV
  Other Names: Bavencio; MSB-0010718C; MSB0010718C
Drug: Berzosertib — Given IV
  Other Names: 2-Pyrazinamine, 3-(3-(4-((Methylamino)methyl)phenyl)-5-isoxazolyl)-5-(4-((1-methylethyl)sulfonyl)phenyl)-; M 6620; M6620; VX 970; VX-970; VX970

SUMMARY:
This phase I/II trial studies the side effects and best dose of avelumab with M6620 in treating patients with deoxyribonucleic acid (DNA) damage repair (DDR) deficient solid tumors that have spread to other places in the body (metastatic) or cannot be removed by surgery (unresectable). DDR deficiency refers to a decrease in the ability of cells to respond to damaged DNA and to repair the damage, which can be caused by genetic mutations. Immunotherapy with monoclonal antibodies, such as avelumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. M6620 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving avelumab together with M6620 may help to control DDR deficient metastatic or unresectable solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of the combination of berzosertib (M6620) and avelumab in patients with DNA damage response (DDR) deficient advanced solid tumors. (Arm A: M6620 + avelumab) II. To establish the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of the combination of M6620 and avelumab in patients with DDR deficient advanced solid tumors. (Arm A: M6620 + avelumab)

SECONDARY OBJECTIVES:

I. To determine the clinical benefit of the combination as defined by clinical benefit rate (CBR) - complete response [CR] + partial response [PR] + stable disease [SD] > 6 months (CR + PR + SD > 6 months). (Arm A: M6620 + avelumab) II. To assess clinical benefit of the combination as defined by objective response rate (ORR), overall survival (OS), duration of response (DoR) and progression free survival (PFS). (Arm A: M6620 + avelumab)

EXPLORATORY OBJECTIVES:

I. To evaluate clinical benefit of the combination of M6620 and avelumab based on specific DDR aberrations. (Arm A: M6620 + avelumab) II. To evaluate clinical benefit of the combination of M6620 and avelumab based on DDR gene expression signatures. (Arm A: M6620 + avelumab) III. To evaluate the impact of treatment on programmed death ligand 1 (PD-L1) expression and immune cell populations. (Arm A: M6620 + avelumab) IV. To assess potential mechanisms of resistance by comparing pre- and on-treatment biopsies in responders and non-responders. (Arm A: M6620 + avelumab) V. To evaluate the pharmacokinetic (PK) and pharmacodynamic (PD) profile of M6620 in combination with avelumab in patients with DDR deficient advanced solid tumors. (Arm A: M6620 + avelumab)

OUTLINE: This is a phase I, dose-escalation study of M6620, followed by a phase II study.

Patients receive avelumab intravenously (IV) over 60 minutes on days 1 and 15, and M6620 IV over 60 minutes on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30, 60, and 90 days, then every 12 weeks afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative measures do not exist or are no longer effective
* Subjects will be eligible for this study based on the presence of actionable aberrations in one or more of the following DNA damage response (DDR) genes: ARID1A, ATM, ATR, ATRX, BAP1, BARD1, BRCA1/2, BRIP1, CDK12, CHEK2, FANCA, FANCC, FANCD2, FANCE, FANCF, FANCM, MRE11A, MSH2, NBN (NBS1), PALB2, RAD51, RAD51C, RAD51D, SMARCB1, and VHL, or other related genes at the discretion of the principal investigator in consultation with the MD Anderson Cancer Center Institute for Personalized Cancer Therapy Precision Oncology Decision Support (PODS) group. Variant interpretation for actionability will be performed by PODS
* Subjects with germline defects in DDR genes are eligible for this trial
* The collection of archival tumor tissue (within 1 year prior to study enrollment) will be mandatory. Tumor biopsies on cycle 1 day 15 will be mandatory. Subjects will not be put at undue risk to obtain the biopsy at cycle 1 day 15 (C1D15). A biopsy at C1D15 will not be required if it poses a serious/severe complication risk greater than 2%. All other biopsy time points are not mandatory but will be strongly encouraged where feasible. These include at baseline and at disease progression. Archival and fresh tissue requests can be waived in exceptional circumstances with principal investigator (PI) approval and only where rationale is documented
* Subjects must have received at least 1 line of systemic therapy in the advanced/metastatic setting. Subjects with diseases without known effective options, and subjects who had declined standard of care therapy prior to study introduction are also eligible
* Subjects enrolling in the dose escalation should have progressed on or be intolerant to all therapies known to confer a clinical benefit. Subjects must not have refused all available therapies
* Subjects who have received prior therapy with immune checkpoint inhibitors (ICIs) are eligible for this trial. Subjects with a standard-of-care option for an immune checkpoint inhibitor are eligible
* Subjects must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1, or patients may have bone metastatic disease evaluable by Prostate Cancer Working Group 3 (PCWG3) for subjects with metastatic castration-resistant prostate cancer (CRPC), or according to tumor evaluation criteria best suited and accepted for the tumor type to be evaluated
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Subjects must have a life expectancy >= 12 weeks
* Absolute neutrophil count >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L
* Total bilirubin =< 1.5 X the institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/ alanine aminotransferase (ALT) serum glutamic-pyruvic transaminase (SGPT) =< 2.5 X institutional ULN or =< 5 X institutional ULN in the presence of liver metastases
* Serum creatinine =< 2 X ULN or estimated creatinine clearance >= 30 mL/min according to the Cockcroft-Gault formula
* Female patients of childbearing potential must have a negative serum or urine pregnancy test at screening (and again at baseline just prior to first administration of study drugs)
* Female patients of non-childbearing potential must meet at least 1 of the following criteria:

  * Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months, with no alternative pathological or physiological cause;
  * Have undergone a documented hysterectomy and/or bilateral oophorectomy
  * Have medically confirmed ovarian failure All other female patients (including female patients with tubal ligation) are considered to be of childbearing potential
* Women of childbearing potential and fertile men must agree to use adequate contraception when sexually active from signing of the informed consent form for the full study until at least 6 months after the last study drug administration. Patients must agree to utilize 2 reliable and acceptable methods of contraception simultaneously. A man is considered fertile after puberty unless permanently sterile by bilateral orchiectomy. Men taking part in this study are advised not to father a child during and up to 6 months after treatment; prior to treatment, advice should be sought for conserving sperm due to the chance of irreversible infertility as a consequence of treatment. Female partners of childbearing potential from male study patients have to use adequate contraception / birth control between signing of the informed consent and 6 months after the last administration of the study drug if the male study patient is not sterilized. The investigator or a designated associate is requested to advise the patient how to achieve highly effective birth control. Highly effective (failure rate of less than 1% per year) contraception methods, when used consistently and correctly, include:

  * Combined (estrogen and progestin containing: oral, intravaginal, transdermal) and progestin-only (oral, injectable, implantable) hormonal contraception associated with inhibition of ovulation
  * Intra-uterine device or intrauterine hormone-releasing system
  * Bilateral tubal occlusion or vasectomized partner (provided that partner is the sole sexual partner and has received medical assessment of the surgical success)
  * Sexual abstinence (reliability to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient) Male patients with a female partner of reproductive potential must use a condom and ensure that an additional form of contraception is also used during treatment and until 6 months after last study drug administration. Patients must agree to utilize 2 reliable and acceptable methods of contraception simultaneously
* Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other procedures
* Human immunodeficiency virus (HIV)-infected (HIV1/2 antibody-positive) patients may participate IF they meet all the following eligibility requirements:

  * They must be on an anti-retroviral regimen with evidence of at least two undetectable viral loads within the past 6 months on this same regimen; the most recent undetectable viral load must be within the past 12 weeks
  * They must have a CD4 count >= 250 cells/mcL over the past 6 months on this same anti-retroviral regimen and must not have had a CD4 count < 200 cells/ mcL over the past 2 years, unless it was deemed related to the cancer and/or chemotherapy-induced bone marrow suppression

    * For patients who have received chemotherapy in the past 6 months, a CD4 count < 250 cells/mcL during chemotherapy is permitted as long as viral loads were undetectable during this same chemotherapy
  * They must have an undetectable viral load and a CD4 count >= 250 cells/mcL within 7 days of enrolment
  * They must not be currently receiving prophylactic therapy for an opportunistic infection and must not have had an opportunistic infection within the past 6 months

Exclusion Criteria:

* Anticancer systemic therapy or radiotherapy within 4 weeks or 5 half-lives, whichever is shorter prior to starting the study agents. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided it has been completed 2 weeks prior to study enrollment, and no clinically significant toxicities are expected (e.g., mucositis, esophagitis)
* Known symptomatic brain metastases requiring steroids. Patients with previously treated diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to study enrollment, have discontinued corticosteroid treatment for these metastases for at least 4 weeks and are neurologically stable
* Current use of immunosuppressive medication at the time of study enrollment, EXCEPT for the following permitted steroids:

  * Intranasal, inhaled, topical steroids, eye drops, or local steroid injection (e.g., intra-articular injection)
  * Systemic corticosteroids at physiologic doses =< 10 mg/day of prednisone or equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g. computed tomography [CT] scan premedication)
* Subjects who had major surgery within 4 weeks prior to study enrollment
* Known prior severe hypersensitivity to investigational products or any component in their formulations, including known severe hypersensitivity reactions to monoclonal antibodies (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version [v] 5 grade >= 3)
* Active infection requiring systemic therapy
* Known history of immune-mediated colitis, inflammatory bowel disease, pneumonitis, and pulmonary fibrosis
* Active or prior autoimmune disease that may deteriorate when receiving an immunostimulatory agent. Patients with type I diabetes, vitiligo, psoriasis, or hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible
* Prior organ transplantation including allogenic stem cell transplantation
* Diagnosis of myelodysplastic syndrome (MDS)
* Vaccination within 4 weeks of study enrollment and while on trial is prohibited except for the administration of inactivated vaccines
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 month prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (>= New York Heart Association Classification class II) or a serious cardiac arrhythmia requiring medication
* Other acute or chronic medical or psychiatric conditions including but not limited to recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results, and in the judgement of the Investigator, would make the patient inappropriate for entry into this study
* Pregnant female patients, breastfeeding female patients, fertile male patients, and female patients of childbearing potential who are unwilling or unable to use 2 highly effective methods of contraception as outlined in this protocol for the duration of the study, and for at least 6 months after the last dose of study drug administration
* Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV ribonucleic acid (RNA) if anti-HCV antibody screening test is positive)
* Known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ bladder cancer, or other cancer for which the patient has been disease-free for >= 2 years
* Persisting toxicity related to prior therapy (NCI CTCAE v5 grade > 1); however, alopecia and sensory neuropathy grade =< 2, or other grade =< 2 AEs not constituting a safety risk, based on the investigator's judgement, are acceptable
* Subjects receiving treatment with strong inhibitors or inducers of CYP3A4 that cannot be discontinued before start of investigational treatment and for the duration of study
* Subjects with ongoing toxicity (any grade) and/or resolved ICI toxicity (grade 3 or higher only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A Yap, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A phase I/II single center study performed at MD Anderson Cancer Center. Patients were eligible if they had (1) advanced solid tumors for hiwch curative measures did not exist or were not longer effective and (2) had actionable mutations in DNA Damage Response (DDR) genes (ARID1A, ATM, ATR, ATRX, BAP1, BARD1, BRCA1/2, BRIP1, CDK12, CHEK2, FANCA, FANCC, FANCD2, FANCE, FANCF, FANCM, MRE11A, MSH2, NBN (NBS1), PALB2, RAD51, RAD51C, RAD51D, SMARCB1, and VHL).
Pre-assignment Details: Patients were first enrolled in dose escalation cohorts to determine the recommendated phase 2 dose before enrolling patients into dose expansion cohorts.
Period: Overall Study
Arm/Group | Escalation Dose Level 1 | Escalation Dose Level 2 | Expansion Dose Level 1 | Expansion Dose Level 2
Started | 7 | 6 | 0 | 10
Completed | 0 | 0 | 0 | 0
Not Completed | 7 | 6 | 0 | 10
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Progression | 6 | 6 | 0 | 10

BASELINE CHARACTERISTICS:
Population: 23 patients were treated across 3 study cohorts. No patients were treated in the Expansion Dose Level 1 cohort.
Groups:
- Total: Total of all reporting groups
Arm/Group | Escalation Dose Level 1 | Escalation Dose Level 2 | Expansion Dose Level 1 | Expansion Dose Level 2 | Total
Number analyzed (Participants) | 7 | 6 | 0 | 10 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  | 0 | 0
  Between 18 and 65 years | 2 | 6 |  | 7 | 15
  >=65 years | 5 | 0 |  | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 |  | 3 | 12
  Male | 2 | 2 |  | 7 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 |  | 3 | 4
  Not Hispanic or Latino | 6 | 6 |  | 7 | 19
  Unknown or Not Reported | 0 | 0 |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0 | 0
  Asian | 1 | 1 |  | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0 | 0
  Black or African American | 0 | 0 |  | 0 | 0
  White | 6 | 4 |  | 10 | 20
  More than one race | 0 | 0 |  | 0 | 0
  Unknown or Not Reported | 0 | 1 |  | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 |  | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose Limiting Toxicities (DLT) as a Measure of Safety Profile to Determine the Recommended Phase 2 Dose (RP2D).
Description: A DLT was evaluated according to the NCI CTCAE 5.0 & defined as: grade 4 neutropenia lasting greater than 7 days or febrile neutropenia, grade 3 thrombocytopenia with bleeding or grade 4 thrombocytopenia lasting greater than 7 days, any treatment related adverse event that in the opinion of the safety monitoring committee exposes participants to unacceptable risk, a delay of more than 4 weeks before receiving the next scheduled study drug due to persisting toxicities attributable to study drugs, grade 3 nausea, vomiting or diarrhea lasting greater than 72 hours with optimal care, grade 3 fatigue lasting greater or equal to 7 days, grade 3 pneumonitis of any duration, any grade 4 immune related toxicities, any other grade 3 or greater non-hematological AE, including infusion-related reactions of any duration, liver enzymes greater than 3 times above the upper limit of normal and concurrent total bilirubin elevation that is greater than 2 times above the upper limit of normal.
Time Frame: The DLT monitoring time frame was the first 28-days of study participation (Cycle 1).
Population: To be evaluable for DLT, patients must have received >75% of the planned dose of the investigational products in the combination during Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation Dose Level 1 | Escalation Dose Level 2 | Expansion Dose Level 1 | Expansion Dose Level 2
Number analyzed (Participants) | 7 | 6 | 0 | 10
Participants
  DLT | 1 | 0 |  | 0
  Not DLT | 5 | 6 |  | 10
  Not evaluable for DLT | 1 | 0 |  | 0

ADVERSE EVENTS:
Time Frame: Approximately three years and four months, from the time the first patient signed the informed consent, through the treatment period, and up to 90 days after the last administration of the lst dose of study drug.
Description: Adverse events (AEs) were graded based on the Common Terminology Criteria for Adverse Events (CTCAE) Version 5. All adverse events were captured from the time of signing consent through 90 days after the last dose of study drug, until all drug related toxicities have resolved, or 30 days prior to initiating a new anticancer therapy, whichever occurred first.
Arm/Group | Escalation Dose Level 1 | Escalation Dose Level 2 | Expansion Dose Level 1 | Expansion Dose Level 2
All-Cause Mortality (participants affected / at risk) | 6/7 | 4/6 | 0/0 | 7/10
Serious Adverse Events (participants affected / at risk) | 2/7 | 2/6 | 0/0 | 4/10
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 0/0 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Escalation Dose Level 1 (N=7) | Escalation Dose Level 2 (N=6) | Expansion Dose Level 1 (N=0) | Expansion Dose Level 2 (N=10)
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lung Infection (Infections and infestations) | 1 | 0 | 0 | 0
Disease Progression (General disorders) | 0 | 1 | 0 | 0
Small Intestinal obstruction (Infections and infestations) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Tumor pain (General disorders) | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | NA | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Escalation Dose Level 1 (N=7) | Escalation Dose Level 2 (N=6) | Expansion Dose Level 1 (N=0) | Expansion Dose Level 2 (N=10)
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 4 | 3 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 4 | 0 | 3
Anorexia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 4 | 2 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bloating (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 2
Chills (General disorders) | 2 | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Creatinine increased (Investigations) | 3 | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 3 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 4
Eye disorders (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 2
Fever (General disorders) | 3 | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Follicular Lymphoma (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Gait Disturbance (General disorders) | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 2
Hematuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hyperurocemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0
Hypothyroidism (General disorders) | 1 | 0 | 0 | 0
Infusion related reaction (General disorders) | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 1 | 0 | 0 | 1
lung infection (Infections and infestations) | 0 | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Neutrophil count decreased (Investigations) | 2 | 2 | 0 | 1
non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0
Pain (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
platelet count decreased (Investigations) | 2 | 0 | 0 | 5
Pruitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
serum amylase increased (Investigations) | 2 | 0 | 0 | 0
sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0 | 1
Weight loss (Investigations) | 0 | 1 | 0 | 0
White blood cell decreased (Investigations) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT04266912/Prot_SAP_000.pdf